CLINICAL TRIAL: NCT02787603
Title: Evaluation of Procalcitonin in the Early Antibiotic Therapy Interruption in Patient With Bacterial Pulmonary infeCtion and Decompensated Acute Heart Failure
Brief Title: Procalcitonin in Early Antibiotic Interruption in Patient With Bacterial Pulmonary infeCtion and Acute Heart Failure
Acronym: EPICAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSInCor-Procalcitonin Clinical
Record Dates: First submitted 2016-05-25; First posted 2016-06-01 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-01

CONDITIONS: Respiratory Tract Infections; Pneumonia, Bacterial; Heart Failure
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia, Bacterial; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Experimental): Interruption of antibiotic treatment due to PCT measurement
  Interventions: Other: Interruption of antibiotic treatment due to PCT measurement
- group B (No Intervention): Antibiotic therapy period will be determined by the physician without the knowledge of PCT levels.

INTERVENTIONS:
Other: Interruption of antibiotic treatment due to PCT measurement — In group A at day 5, if the patient shows no clinical signs of infection and PCT levels < 0,25ng/mL OR PCT > 0,25 ng/mL AND 80% reduction in comparison with day 0 PCT levels, antibiotic will be interrupted. If there is a constant level or decrease less than 80% when compared day 0 or 5, there is no change in antibiotic treatment.
  Arms: group A

SUMMARY:
Introduction: Acute Heart Failure is frequently decompensated by pulmonary infection, but the diagnosis of pulmonary infection sometimes is difficult in these patients due to similar signals and clinical symptoms in both pathologies. Furthermore, when it is possible the diagnosis of pulmonary infection, physicians may have difficult to determine etiology and delaying antibiotic therapy. Procalcitonin (PCT) have been used like a biomarker to determine the period of use of antibiotics in patients with acute respiratory infections. It is specific for bacterial infections and it have showed as a marker of severity infection and may help to determine interruption period of antibiotic therapy in a safety way for the patient. Aim: Evaluate levels of PCT related to interruption of antibiotics in patients with decompensated acute heart failure (DAHF) with suspected bacterial pulmonary infection. Methods: In this pilot project will be included around 100 patients, randomized in two groups: group A (PCT levels may guide the interruption of antibiotic at day 5) or group B (antibiotic period will be determined by the physician without the knowledge of PCT levels). Will be collected laboratorial and clinical data at days 0,3 and 5. Both groups will be compared to evaluate PCT levels and total period of antibiotic therapy, hospitalization and readmission in 30 days. This study will determine the sensibility/specificity of PCT in patients with DAHF.

DETAILED DESCRIPTION:
It is a single-center study, randomized, controlled, prospective cohort and interventional not blind. DAHF diagnosis will consider symptoms, physical examination, x ray and other image methods and BNP ou NTproBNP levels. Pulmonary infection diagnosis will "Infectious Disease Society of America / American Thoracic Society Consensus Guidelines on the Management of Community-Acquired Pneumonia in Adults" criteria, that include fever, cough, sputum, pleuritic pain, positive pulmonary image and physical examination. PCT and NTproBNP levels will be measured in miniVIDAS® (bioMérieux Clinical Diagnostics, France). Statistics includes descriptive analysis. Parametric data will be evaluated using T test and non parametric data with Mann-Whitney-Wilcoxon test. Multivariative analysis related to diagnosis, mortality and morbidity will be performed by Cox regression model. Sensibility and specificity will be calculated by ROC curve. Statistical significancy will be considered when p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* DAHF diagnosis and suspected pulmonary infection
* BNP ≥ 500 pg/mL or NTproBNP ≥ 450 pg/mL for patients until 50 years old.
* BNP ≥ 500 pg/mL or NTproBNP ≥ 900 pg/mL for patients with 51 - 75 years old.
* BNP ≥ 500 pg/mL or NTproBNP ≥ 1800 pg/mL for patients older than 75 years.

Exclusion Criteria:

* Antibiotic use (oral or endovenous) in the last 15 days;
* Acute coronary syndrome;
* Creatinine > 3,0 mg/dL or hemodialysis;
* Pregnancy;
* Second suspectec infection;
* Suspected pulmonary thromboembolism;
* cancer;
* myocarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Total period of antibiotic therapy | 30 days

SECONDARY OUTCOMES:
hospitalization | 30 days
mortality | 30 days
PCT levels during antibiotic therapy | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Mucio Tavares, PhD MD, Principal Investigator — Unidade Clínica de Emergência
Locations (1):
- Unidade Clínica de Emergência - Instituto do Coração InCor HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Maisel A, Neath SX, Landsberg J, Mueller C, Nowak RM, Peacock WF, Ponikowski P, Mockel M, Hogan C, Wu AH, Richards M, Clopton P, Filippatos GS, Di Somma S, Anand I, Ng LL, Daniels LB, Christenson RH, Potocki M, McCord J, Terracciano G, Hartmann O, Bergmann A, Morgenthaler NG, Anker SD. Use of procalcitonin for the diagnosis of pneumonia in patients presenting with a chief complaint of dyspnoea: results from the BACH (Biomarkers in Acute Heart Failure) trial. Eur J Heart Fail. 2012 Mar;14(3):278-86. doi: 10.1093/eurjhf/hfr177. Epub 2012 Feb 2. PMID 22302662
- [Result] Schuetz P, Albrich W, Mueller B. Procalcitonin for diagnosis of infection and guide to antibiotic decisions: past, present and future. BMC Med. 2011 Sep 22;9:107. doi: 10.1186/1741-7015-9-107. PMID 21936959
- [Result] Bafadhel M, Clark TW, Reid C, Medina MJ, Batham S, Barer MR, Nicholson KG, Brightling CE. Procalcitonin and C-reactive protein in hospitalized adult patients with community-acquired pneumonia or exacerbation of asthma or COPD. Chest. 2011 Jun;139(6):1410-1418. doi: 10.1378/chest.10-1747. Epub 2010 Oct 28. PMID 21030489
- [Result] Bouadma L, Luyt CE, Tubach F, Cracco C, Alvarez A, Schwebel C, Schortgen F, Lasocki S, Veber B, Dehoux M, Bernard M, Pasquet B, Regnier B, Brun-Buisson C, Chastre J, Wolff M; PRORATA trial group. Use of procalcitonin to reduce patients' exposure to antibiotics in intensive care units (PRORATA trial): a multicentre randomised controlled trial. Lancet. 2010 Feb 6;375(9713):463-74. doi: 10.1016/S0140-6736(09)61879-1. Epub 2010 Jan 25. PMID 20097417
- [Result] Schuetz P, Kutz A, Grolimund E, Haubitz S, Demann D, Vogeli A, Hitz F, Christ-Crain M, Thomann R, Falconnier C, Hoess C, Henzen C, Marlowe RJ, Zimmerli W, Mueller B; ProHOSP Study Group. Excluding infection through procalcitonin testing improves outcomes of congestive heart failure patients presenting with acute respiratory symptoms: results from the randomized ProHOSP trial. Int J Cardiol. 2014 Aug 20;175(3):464-72. doi: 10.1016/j.ijcard.2014.06.022. Epub 2014 Jun 27. PMID 25005339